CLINICAL TRIAL: NCT01823978
Title: A Phase I Study of BPX-201 Vaccine Plus AP1903 in Patients With Metastatic Castrate Resistant Prostate Cancer (mCRPC)
Brief Title: Safety Study of BPX-201 Dendritic Cell Vaccine Plus AP1903 in Metastatic Castrate Resistent Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-PC-002
Record Dates: First submitted 2013-03-21; First posted 2013-04-04 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2018-11

CONDITIONS: Castrate Resistent Prostate Cancer
Keywords: metastatic; castration resistant prostate cancer; Therapeutic Vaccine; Dendritic cell; BPX-201; BPX201; AP1903
MeSH Terms: conditions — Neoplasm Metastasis | interventions — AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BPX-201 (Experimental): BPX-201 vaccine plus AP1903
  Interventions: Biological: BPX-201 vaccine plus AP1903

INTERVENTIONS:
Biological: BPX-201 vaccine plus AP1903 — The trial design consists of 3 cohorts of 6 patients each, receiving escalating doses of BPX-201 of 10 million (M), 20M and 40M cells, respectively. Dose escalation will occur according to a 3+3 design. Patients will receive administration of BPX-201 every other week for 6 cycles (1 cycle equals 2 weeks). Approximately 1.6 mL of BPX-201 will be administered as 8 intradermal injections (200μL each) at each treatment visit. On the day following each vaccination, a single 40 mg dose of the activating agent, AP1903, will be administered via intravenous (IV) infusion over 2 hours.

SUMMARY:
This is a Phase I, non-randomized, dose escalation study of the safety, biomarkers, and preliminary efficacy of dendritic cell vaccine, BPX-201, plus activating agent, AP1903, in patients with metastatic castrate resistant prostate cancer.

DETAILED DESCRIPTION:
This is a Phase I study of therapeutic vaccine, BPX-201, plus activating agent, AP1903, in patients with mCRPC. Patients will be screened within 8 weeks prior to first vaccine administration (4 weeks prior to leukapheresis). The trial design consists of 3 cohorts of 6 patients each, receiving escalating doses of BPX-201 of 10 million (M), 20M and 40M cells, respectively. Dose escalation will occur according to a 3+3 design. Patients will receive administration of BPX-201 every other week for 6 cycles (1 cycle equals 2 weeks). Approximately 1.6 mL of BPX-201 will be administered as 8 intradermal injections (200μL each) at each treatment visit. On the day following each vaccination, a single 40 mg dose of the activating agent, AP1903, will be administered via intravenous (IV) infusion over 2 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. 18 years of age or older
3. Histologically confirmed, metastatic prostate cancer (positive bone scan and/or measurable disease on CT scan and/or MRI of the abdomen and pelvis).
4. Progressive disease after androgen deprivation, as defined by Prostate Cancer Working Group 2 and/or Response Evaluation Criteria in Solid Tumors criteria
5. Laboratory requirements:

   * Absolute neutrophil count (ANC) ≥ 1500/μL
   * Bilirubin < 1.5 x ULN
   * Hemoglobin > 8 g/dL
   * PSA > 2 ng/mL
   * Platelets > 100,000/µL
   * AST and ALT < 2.5 x ULN
   * Creatinine clearance ≥ 60mL/min
   * Testosterone < 50 ng/dL
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2 and life expectancy > 12 weeks
7. Patients receiving any other hormonal therapy, including any dose of megestrol acetate (Megace), Proscar (finasteride), any herbal product known to decrease PSA levels (e.g. Saw Palmetto, PC-SPES), or agents such as abiraterone, TAK700, MDV3100 as well as any systemic corticosteroid use, must discontinue the agent for at least four weeks prior to study treatment. Progressive disease as defined above must be documented after discontinuation of any hormonal therapy (with the exception of a LHRH agonist).
8. Prior radiation therapy must be completed > 4 weeks prior to enrollment and the patient must have recovered from all toxicity. Prior radiopharmaceuticals (strontium, samarium) must be completed ≥ 8 weeks prior to enrollment.
9. Because of the unknown potential risk to a gamete and/or developing embryo from these investigational therapies, patients must agree to use adequate contraception (barrier method for males) for the duration of study participation, and for three months after discontinuing therapy.

Exclusion Criteria:

1. Prior chemotherapy for prostate cancer, with the exception of neo-adjuvant chemotherapy, because of the potential effect of chemotherapy on the immune system.
2. Prior sipuleucel-T treatment or investigational immunotherapy.
3. Prostate cancer pain requiring regularly scheduled narcotics.
4. Current treatment with systemic steroid therapy (inhaled/topical steroids are acceptable). Systemic corticosteroids must be discontinued for at least 4 weeks prior to first treatment.
5. Clinically active autoimmune disease.
6. Diagnosis of prostate cancer with neuroendocrine differentiation
7. Known presence of central nervous system metastases, pleural effusions or ascites
8. Medical or psychiatric illness that would, in the opinion of the investigator, preclude participation in the study or the ability of patients to provide informed consent for themselves.
9. Cardiovascular disease that meets one of the following: congestive heart failure (New York Heart Association Class III or IV), active angina pectoris, or recent myocardial infarction (within the last 6 months).
10. Concurrent or prior malignancy except for the following:

    * Adequately treated basal or squamous cell skin cancer
    * Adequately treated stage I or II cancer from which the patient is currently in complete remission
    * Any other cancer from which the patient has been disease-free for 5 years
11. Known HIV or other history of immunodeficiency disorder.
12. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or medical (e.g. infectious) illness.
13. Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of BPX-201 and AP1903 hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
14. Any non-oncology vaccine therapy used for prevention of infectious diseases for up to 1 month before BPX-201

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with adverse events as a measure of safety and tolerability | 2 years
  Safety will be measured through the monitoring of AEs, clinical laboratory parameters (hematology, serum chemistry, and urinalysis), vital sign measurements, and physical examinations.

SECONDARY OUTCOMES:
prostatic specific antigen | 3 months
  Measure PSA response and PSA doubling time as measured from PSA nadir through 12 weeks
Progression free survival | 2 years
  Rate of PFS
Reduction in circulating tumor cells | 2 years
  Change from baseline in number of circulating tumor cells
Response to chemotherapy after vaccine | 2 years
  Response to chemotherapy upon progression

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Fong, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Baylor Charles Sammons Cancer Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No